CLINICAL TRIAL: NCT03747237
Title: Assessment of the Relationship Between Edema Measurement Methods After Impacted Mandibular Third Molar Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Dilek Menziletoglu, Principle Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEU
Record Dates: First submitted 2018-09-21; First posted 2018-11-20 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-11

CONDITIONS: Impacted Third Molar Tooth
Keywords: edema; third molar
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. method, Edema measurement methods (Experimental): The surgeon will measure from three different places on the patient's face with the help of a paper ruler to measure the edema.
  Tragus-Pogonion Tragus-Labial Comissura Angulus Mandible-Latheral Cantus Measurements will be made preoperative, postoperative 2. and 7. days and saved as milimetre.
  Interventions: Other: Edema measurement methods
- 2. method, Edema measurement methods (No Intervention): Patients will be given edema scale.With the help of the edema scale, the patients will be evaluated the edema by themselves. When the patient stand in front of the mirror, they will be assessed the edema on their face. And a value between 0 and 5 will be pointed on the scale postoperative 2. and 7. days.

INTERVENTIONS:
Other: Edema measurement methods — A correlation between the results of the first and second methods will be examined.
  Arms: 1. method, Edema measurement methods

SUMMARY:
The aim of this study is to evaluate the correlation between two point distance measurements performed by surgeon on patients face with foldable ruler, which is the most commonly used method, and the subjective scoring will be done by the patient with the help of the edema scale, for measuring edema.

DETAILED DESCRIPTION:
The patients will be selected among the patients who apply for mandibular impacted third molar extraction to Necmettin Erbakan University, Faculty of Dentistry. A total of 60 patients will be included. All third molar operations will be carried out by the same surgeon in all groups with the same technique.Two methods will be used to evaluate the edema on the face.

1. Method The surgeon will measure from three different places on the patient's face ( two point distance) with the help of a paper ruler.

   * Tragus-Pogonion
   * Tragus-Labial Komissura
   * Angulus Mandibula-Lateral Kantus Measurements will be made preoperative, postoperative 2. and 7. days and saved as milimetre.
2. Method Patients will be given edema scale.With the help of the edema scale, the patients will be evaluated the edema by themselves. When the patient stand in front of the mirror, they will be assessed the edema on their face. And a value between 0 and 4 will be pointed on the scale postoperative 2. and 7. days.

A correlation between the results of the first and second methods will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Impacted mandibular third molar teeth (mesioangular, mucosa and bone retantion)
* Patients with any chronic disease and allergy

Exclusion Criteria:

* Smoking
* Pregnancy or lactation
* pericoronitis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Tragus-pogonion measurement will be made with paper ruler. | Up to 1week
  The measurement will be done on the 2. and 7. postoperative day and preoperative.
Tragus-labial comissura measurement will be made with paper ruler. | Up to 1week
  The measurement will be done on the 2. and 7. postoperative day and preoperative.
Angulus mandible-latheral cantus will be made with paper ruler | Up to 1week
  The measurement will be done on the 2. and 7. postoperative day and preoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoglu, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Karatay, Turkey (Türkiye)